CLINICAL TRIAL: NCT06302192
Title: RED-AKI: Renal Doppler in Acute Kidney Injury. Capability of Intrarenal Venous Flow Doppler (IRVF) to Predict Acute Kidney Injury (AKI) in Critically Ill Patients With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Renal Doppler to Predict Acute Kidney Injury (AKI) in ARDS Patients. (RED-AKI Study)
Acronym: RED-AKI
Status: Not yet recruiting | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Professor, Policlinico Hospital
Other Study IDs: 4302
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Acute Kidney Injury; ARDS, Human
Keywords: Renal Doppler
MeSH Terms: conditions — Acute Kidney Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — on day #1, on day #3, on day #7 and on day #14 any 3 ml of urine and 3 ml of blood will be stocked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ARDS+AKI — according to the clinical practice Reanl doppler and VeXUS score will be performed

SUMMARY:
This is a multicenter international observational prospective cohort study. The main questions it aims to answer are:

* PRIMARY AIM: To describe the capability of IRVF demodulation at diagnosis of ARDS to predict development of AKI within 7 days from the ARDS onset
* SECONDARY AIMS: A)Describe the capability of IRVF demodulation or pattern of IRVF (continuous, pulsatility, biphasic, monophasic) to predict development of AKI within 14 days from the ARDS onset. B) To describe the RD parameters and VexUS in the AKI and no AKI patients over time. C) Describe the impact of invasive mechanical ventilation (IMV) on the intrarenal venous congestion and VexUS., D) Evaluation of effect of CRRT on IRVF pattern, VexUS and parameters. E) Describe the feasibility of renal doppler to assess IRVF in critically ill respiratory patients. F) Evaluate the incidence of AKD and CKD Participants will Adult patients with diagnosis of ARDS admitted to intensive care unit and undergoing invasive mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Critically ill patients admitted to intensive care unit with a diagnosis of ARDS according to Berlino criteria
* Beginning of IMV less than 48 hours or Clinical decision to begin IMV.
* Life expectancy > 24 hours
* Informed consent signed

Exclusion Criteria:

No patient will be excluded from the study because of gender, race, ethnicity, or sexual preference.

* AKI prior to the onset of ARDS
* Chronic respiratory failure due to chronic respiratory diseases
* Chronic renal disease (CKD stage ≥ 2) and any ureteral obstruction. Definition of CKD patient is according to the latest guideline KDIGO
* Chronic Heart Failure
* Chronic liver disease
* Major trauma in the past 3 months
* Major surgery in the past 3 months
* Smoking and Alcohol drinking
* BMI ≥ 35
* Patients needing of VV-ECMO and VA-ECMO
* Beginning of positive pressure ventilation more than 48 hours (invasive or no invasive)
* Life expectancy <24 hours
* Cardio Circulatory Arrest
* Neoplasm in chemotherapy/radiotherapy
* Do Not Resuscitate or Comfort Measures
* Pregnancy at ICU admission
* Refused Informed Consent by the patient or surrogate decision-maker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosis of ARDS admitted to intensive care unit and undergoing invasive mechanical ventilation (IMV).
Sampling Method: Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence | 1st april 2024 - 31st of january 2026
  Cumulative incidence of AKI within 7 days from the ARDS onset in demodulated and no-demodulated group

SECONDARY OUTCOMES:
AKI14 | 1st april 2024 - 31st of january 2026
  ) Incidence of AKI within 14 days from the ARDS onset in patient with and without IRVF demodulated or with different IRVF pattern
AKIstage | 1st april 2024 - 31st of january 2026
  VM, RIhil and RIintra, SI, VexUS values in AKI and no AKI patients and in the different AKI stage
cross talk lung-kidney | 1st april 2024 - 31st of january 2026
  invasive mechanical ventilation parameters (PEEP, Pressure of plateau, driving pressure and static compliance of the respiratory system) values and PaCO2 and PaO2/FiO2 values in the demodulated or in any IRVF pattern (continuous, pulsatility, biphasic and monophasic)
CRRT | 1st april 2024 - 31st of january 2026
  IRVF pattern (continuous, pulsatility, biphasic, monophasic), VM, RIhil and RIintra, IRVFhil, SI and VexUS at the beginning and at the discontinuation of CRRT
incidence of failed exam | 1st april 2024 - 31st of january 2026
  Percentage of exams successfully performed among the total of patients admitted to study
CKD progression | 1st april 2024 - 31st of january 2026
  Incidence of CKD Incidence of CKD Cumulative Incidence of CKD

IPD SHARING:
Plan to Share IPD: Undecided